CLINICAL TRIAL: NCT00175344
Title: Does Scar Tissue Massage Improve Postoperative Pain and Function in Women With Breast Cancer? A Randomized Controlled Study.
Brief Title: Does Scar Massage Improve Postoperative Pain and Function in Women With Breast Cancer?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H03-60011
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; scar massage; breast conserving surgery; scar pain; quality of life; Breast cancer treated with breast conserving surgery with or without axillary dissection or sentinel node sampling.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Arm A: Self-administered massage of the postoperative scar after breast cancer surgery.
  Interventions: Procedure: Scar massage.

INTERVENTIONS:
Procedure: Scar massage. — To objectively evaluate the effects of scar massage, those who agree to participate will be randomly assigned to one of two groups. One group will be taught to perform self-massage of the scars as soon as the scars have adequately healed. The massage should be done about 10 minutes each day for a total of 6 months. The other group will not be taught self-massage and will be asked to not massage their breast scars.

SUMMARY:
All patients undergoing breast cancer surgery are left with scars which can significantly affect their physical and psychological well being. Patients with breast cancer, motivated to optimize healing and function, have inquired about the advisability of scar massage after surgery. Although this is a popular technique advocated by physiotherapists and massage therapists to improve pain, range of motion, and scar pliability, there is currently no scientific research to prove the benefits and/or risks of scar massage in breast cancer patients. We propose to study the effect of scar massage on pain, arm function, scar formation, and quality of life in patients with breast cancer. Patients who have had breast cancer surgery and who have been referred to the BC Cancer Agency, Vancouver Island Centre will be offered participation in this research study. To objectively evaluate the effects of scar massage, those who agree to participate will be randomly assigned to one of two groups. One group will be taught to perform self-massage of the scars as soon as the scars have adequately healed. The massage should be done about 10 minutes each day for a total of 6 months. The other group will not be taught self-massage and will be asked to not massage their breast scars. In both groups, we will monitor pain, upper body range of motion, scar characteristics and quality of life using standardized criteria for 2 years from the time of surgery. Problems with infections or blood or fluid accumulation at the scar areas will also be monitored. After 2 years, the information collected will be analyzed and compared to see if there are differences in pain, function or quality of life between the two groups. The results from this study will provide scientific proof of whether or not scar massage after surgery is beneficial for patients with breast cancer.

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial design. Women who have undergone breast cancer surgery (breast conserving surgery or mastectomy) and who meet the eligibility criteria specified will be offered study participation. After obtaining informed consent, subjects will be randomized between two cohorts: scar massage (intervention group) versus no scar massage (control group). The primary outcome is scar-related pain (scored using the McGill Pain Questionnaire Short Form). The secondary outcomes are: upper body range of motion, physical parameters of the scar (pliability, scar height, vascularity and pigmentation scored using the Vancouver Scar Scale), lymphedema (evaluated by arm circumference measurements) and quality of life (using the Functional Assessment of Cancer Therapy (FACT)-B breast cancer-specific instrument).

A sample size of 143 patients per arm was estimated to detect a 30% difference in the primary outcome of postoperative scar-related pain between the intervention and the control groups with 80% statistical power.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to provide informed consent and be physically able to perform daily self-administered breast scar massage
* Female or male patients with histologically-confirmed invasive or in situ breast cancer
* Definitive surgery with BCS or mastectomy +/- axillary dissection or sentinel node sampling
* Adequate surgical healing as judged by treating oncologist during pre-enrolment assessment
* Age 18 years or older with ability to provide written informed consent.
* Ability to start massage within 8 weeks from surgery and comply with daily regimen if randomized to the intervention cohort
* Ability to comply with not performing massage if randomized to the control cohort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is scar-related pain (scored using the McGill Pain Questionnaire Short Form). | Two years

SECONDARY OUTCOMES:
The secondary outcomes are: upper body range of motion, physical parameters of the scar (pliability, scar height, vascularity and pigmentation scored using the Vancouver Scar Scale), lymphedema (evaluated by arm circumference measurements) and quality of | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Truong, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Cancer Agency - Vancouver Island, Victoria, British Columbia, Canada